CLINICAL TRIAL: NCT05412303
Title: Vaso-inotropic Score and ECMO-VA Support in Post-cardiotomy Cardiogenic Shock.
Acronym: ECMOVIS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GUINOT 2022
Record Dates: First submitted 2022-05-23; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: EMCO-VA
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With ECMO-VA: postcardiotomy cardiogenic shosck supported by ECMO-VA
  Interventions: Other: data collection
- Without ECMO-VA: Post cardiotomy cardiogenic shock medically treated (inotrope and vasopressor)
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — age, gender, body weight, height, personal medical history, ASA score, EuroSCORE2, type of cardiac surgery, the preoperative left ventricular ejection fraction, the duration of CPB, the duration of aortic clamping, the need for intraoperative blood transfusion, norepinephrine, dobutamine, creatinine value, time to extubation (hours), any occurrence of complications during the stay in the ICU or in the hospital, and the LOS in the ICU and hospital

SUMMARY:
Veno-arterial extracorporeal membrane oxygenation (VA-ECMO) is a well-established lifesaving treatment for refractory cardiogenic shock, with or without concomitant respiratory failure. VA-ECMO is usually started in presence of refractory low cardiac output syndrome following CPB weaning. Currently, there is no consensus about the best timing for implantation and initiation of VA-ECMO in this setting. Some publications have suggested that VIS score could be used to determine the necessity of VA-ECMO in cardiologic area. It was demonstrated that a VIS score between 20 and 40 may be a cut-off value to discuss the implantation of VA-ECMO. Post cardiotomy shock is a very interesting setting because the timing of cardiogenic shock is known and several bias are more controlled than in medical area.

Based on the well-established ability of VIS Score in predicting mortality, we will investigate the role of the VIS Score as a determinant for early VA-ECMO implantation in patients suffering of post-cardiotomy cardiogenic shock.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* Cardiac surgery with cardiopulmonary bypass
* Post cardiotomy cardiogenic shock
* ECMO-VA implanted in OR

Exclusion Criteria:

* LVAD
* Heart transplantation
* Incomplete data in relation to outcomes
* Cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post cardiotomy cardiogenic shock
Sampling Method: Non-Probability Sample
Enrollment: 2769 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Pourcentage of death | Day 30

SECONDARY OUTCOMES:
1 - Number of complications | Day 30
  1- cardiac, neurological, renal, respiratory, red blood transfusion complication
2 - number of days in intensive care | through study completion, up to 15 days
3 - number of days in hospital | through study completion, up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France